CLINICAL TRIAL: NCT01457794
Title: OPUS(Optimal Well-being, Development and Health for Danish Children Through a Healthy New Nordic Diet) School Meal Study
Brief Title: OPUS School Meal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arne Astrup (Other)
Collaborators: Technical University of Denmark (Other); University of Aarhus (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Arne Astrup, Professor, MD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D208; H-1-2010-124 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome X; Fatty Acids, Omega-3; Learning; Attention; Nutritional Status; Nutrition Assessments; Body Weight; Physical Activity; Sleep; Child Nutrition Sciences
MeSH Terms: conditions — Metabolic Syndrome; Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NewNordicDiet first (Other): Intervention with NND for 3 mo then no intervention for 3 mo
  Interventions: Other: School meals based on the principles of the New Nordic Diet
- NewNordicDiet last (Other): No intervention for 3 mo and then intervention with NND for 3 mo
  Interventions: Other: School meals based on the principles of the New Nordic Diet

INTERVENTIONS:
Other: School meals based on the principles of the New Nordic Diet — The study participants are provided with three daily school meals for 3 month

SUMMARY:
The aim of this randomized crossover study, is to investigate the effect of school meals based on a sustainable New Nordic Diet on growth, learning abilities, well-being, sleep quality, physical activity and risk markers of cardiovascular disease (CVD), type II diabetes and osteoporosis in 8-11 year old Danish school children.

The participating 3rd and 4th grades on 9 selected primary schools will be randomized to either start receiving New Nordic Diet school meals for 3 month(mo) or to eat their habitual school lunch for 3 mo and then crossover for additional 3 mo. All participants will be examined three times; at baseline, after 3 mo and after 6 mo.

ELIGIBILITY:
Inclusion Criteria:

* Pupils in 3rd and 4th grades
* Primary Schools in the Zealand Region and Capital Region of Denmark
* Schools with an available school kitchen, that can be approved by the food authorities
* Schools where at least 60 % of the pupils in three or more classes signs up to participate in the Study

Exclusion Criteria:

* The children should not participate in a scientific study or have participated in a scientific study within the last 4 weeks. This, however depends on the character of the other study.
* The children must not suffer from serious food allergies or food intolerance.
* The children must not suffer from diseases or conditions that makes them ill-suited for participation in the study, eg. malabsorptive conditions or serious mental disorders
* The Schools must not offer an well-established common meal plan, that provides most of the pupils with healthy food on a daily basis

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 834 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome score | Change during 3 month of intervention compared with change during 3 month control period
  The metabolic syndrome score is a continuous z-score based on individual z-scores for waist circumference (WC), mean arterial pressure (MAP), serum high density lipoprotein (HDL), Serum triglyceride (TG) and Homeostasis Model Assessment (HOMA) index. It´s an internal score meaning that the basis for the score is the distribution of values in this study population at baseline.
Concentration Performance | Change during 3 month of intervention compared with change during 3 month control period
  Concentration Performance is assessed by means of a concentration test called the D2-test of Attention. Concentration Performance is derived from the number of correctly crossed out relevant items minus the errors of commission (confused).

SECONDARY OUTCOMES:
Early Cardiovascular Risk Markers | Change during 3 month of intervention compared with change during 3 month control period
  Systolic and diastolic blood pressure, serum blood cholesterol (total, Low Density Lipoprotein (LDL), Very Low Density Lipoprotein (VLDL) and HDL) and TG, plasma glucose, serum insulin and the HOMA index.
Other metabolic syndrome scores | Change during 3 month of intervention compared with change during 3 month control period
  Other metabolic syndrome scores will be calculated as continuous z-scores based on each of the individual z-scores for Waist Circumference (WC), Mean Arterial Pressure (MAP), serum High Density Lipoprotein (HDL), serum Triglyceride (TG) and insulin, separately, and possibly with weighted contribution of each of the risk markers to the score.
Inflammatory markers | Change during 3 month of intervention compared with change during 3 month control period
  Plasma concentrations of the cytokines Interleucin-6 (IL-6) and Tumor Necrosis Factor (TNF) alfa, the adipokine adiponectin and the acute-phase protein c-reactive protein (CRP) (measured as high-sensitive) in plasma will be used as markers of subclinical inflammation and related to the other early metabolic syndrome and cardiovascular risk markers.
Illnesses and use of medicine | Change during 3 month of intervention compared with change during 3 month control period
  Self-reported data collected by computer-assisted questionnaire interview with the parents, either personal (month 0) or by telephone (month 3 and 6). Outcomes are the number of days, during the last two weeks, with: asthma symptoms, use of asthma-medicine, hay-fever symptoms, use of hay-fever-medicine, atopic eczema, symptoms such as sore throat or fever, and the use of pain killers or antibiotics. The number of days of absence from school due to illness, the number of days of illness during weekends and holidays, and number of visits to the doctor will also be evaluated.
Use of ADHD medicine | Change during 3 month of intervention compared with change during 3 month control period
  Among those children with a diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) or Attention Deficit Disorder (ADD), the mean daily dose of methylphenidate (based on reported intake of drugs containing this substance) during the last two weeks will be evaluated.
General fatty acid composition of whole-blood | Change during 3 month of intervention compared with change during 3 month control period
  Content of saturated fatty acids, monounsaturated fatty acids, polyunsaturated fatty acids, total n-3 and n-6 polyunsaturated fatty acids and the n-6:n-3 ratio in whole-blood measured as weight% relative to the weight of total fatty acids.
Reading proficiency | Change during 3 month of intervention compared with change during 3 month control period
  Reading proficiency is assessed by means of the Danish Sentence Reading test 2 having two measures: Percentage of correct sentences read within eight minutes. Reading speed - number of sentences reached.
Mathematics proficiency | Change during 3 month of intervention compared with change during 3 month control period
  Mathematics proficiency is assessed by means of the Danish MG test for 3rd and 4th grade. They each have one measure: Number of correct results within 45 minutes.
Learning | Change during 3 month of intervention compared with change during 3 month control period
  Student learning is assessed by means of the Danish LRS Learning Rating Scale filled out by students. The scale contains four subscales and one combined scale (sum score) adding the four subscales. The subscales cover: academic learning, social situation in school, teaching style appropriateness, and school expectations.
Wellness | Change during 3 month of intervention compared with change during 3 month control period
  Student wellness is assessed by means of the Danish WRS Wellness Rating Scale filled out by students. The scale contains five subscales and one combined scale (sum score) adding the five subscales. The subscales cover: Living environment, school, school mates, family, and self concept.
Physical activity | Change during 3 month of intervention compared with change during 3 month control period
  Physical activity is measured using actigraphy. Outcome measures will be counts/min, time spent in sedentary, light, moderate and vigorous activities.
  Questions regarding TV-watching, playing with videogames and physical activity, will help identify activity-pattern.
Sleep | Change during 3 month of intervention compared with change during 3 month control period
  Sleep is measured using actigraphy with the monitor placed on the right hip for all students and on the non-dominant wrist for a sub-sample. Using a sleep diary, total sleep time and sleep efficiency will be derived from these actigraphy measurements.
  In addition, at month 0, the abbreviated version of the Children's Sleep Habits Questionnaire (CSHQ) is used to identify sleep problems.
Fitness | Change during 3 month of intervention compared with change during 3 month control period
  Fitness is measured using the Andersen test, which is an intermittent running test to estimate maximal oxygen uptake (mL*min-1*kg-1).
Dietary intake | Change during 3 month of intervention compared with change during 3 month control period
  Dietary intake is measured as micro-and macronutrients as well as food groups (e.g. fish and fruit/vegetables) by means of a 7-day dietary survey, which is a web based recall record method developed especially for children. Families without internet access can use a paper version of a 7-day dietary survey. The meal time perception is measured as well.
Body weight and body mass index (BMI) | Change during 3 month of intervention compared with change during 3 month control period
  Body weight (in kg, BMI and BMI z-score calculated on the basis of the current references from the World Health Organization (WHO)
Body composition | Change during 3 month of intervention compared with change during 3 month control period
  Body composition will be determined by Dual energy X-ray Absorptiometry (DXA) scanning. The parameters included are total body Fat Free Mass Index (FFMI in kg/m2), total body Fat Mass Index (FMI in kg/m2), total body fat percentage and the ratio between android and gynoid fat mass in kg.
Appetite-regulating hormones | Change during 3 month of intervention compared with change during 3 month control period
  Leptin and ghrelin. If resources are available at the end of the study period, ghrelin will be separated in acylated and deacylated ghrelin, and both the effect of the intervention on total, acylated, deacylated and the ratio between acylated:deacylated ghrelin will be assessed. If the resources are too tight at the end of the study, only total ghrelin will be used.
Vitamin D status | Baseline and change during 3 month of intervention compared with change during 3 month control period
  Serum concentrations of 25-hydroxyvitamin D [25(OH)D] will be used as marker of vitamin D status, related to food intake and time of season.
Bone Health | Change during 3 month of intervention compared with change during 3 month control period
  Bone Health will be evaluated by DXA scanning (total body and spine Bone Mineral Content (BMC), Bone Mineral Density (BMD), and Bone Area (BA). Osteocalcin and serum Parathyreoideahormon (PTH) are also included as markers of bone health.
General fatty acid composition in whole-blood | Change during 3 month intervnetion compared with change during 3 month control period
Iron status | Change during 3 month intervention compared with 3 month control period
  Whole-blood hemoglobin and serum ferritin will be used as measures of iron status
Attention - other measures | Change during 3 month of intervention compared with change during 3 month control period
  The following five measures from the attention test D2 will be used:
  TN=Total Number of items processed E%=Percentage of errors
Omega-3 index in whole-blood | Change during 3 month of intervention compared with change during 3 month control period
  The Omega-3 index in whole-blood is defined as the weight percentage of eicosapentaenoicacid + the weight percentage of docosahexaenoic acid in whole-blood

OTHER OUTCOMES:
Genotyping | Baseline
  SNPs in genes related to metabolic pathways, messenger molecules, receptors or other genes that may affect efficacy measures in OPUS School Food Project

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Lauritzen L, Sorensen LB, Harslof LB, Ritz C, Stark KD, Astrup A, Dyssegaard CB, Egelund N, Michaelsen KF, Damsgaard CT. Mendelian randomization shows sex-specific associations between long-chain PUFA-related genotypes and cognitive performance in Danish schoolchildren. Am J Clin Nutr. 2017 Jul;106(1):88-95. doi: 10.3945/ajcn.117.152595. Epub 2017 May 17. PMID 28515069
- [Derived] Biltoft-Jensen A, Damsgaard CT, Andersen EW, Ygil KH, Andersen R, Ege M, Christensen T, Thorsen AV, Tetens I, Wu H, Landberg R. Validation of Reported Whole-Grain Intake from a Web-Based Dietary Record against Plasma Alkylresorcinol Concentrations in 8- to 11-Year-Olds Participating in a Randomized Controlled Trial. J Nutr. 2016 Feb;146(2):377-83. doi: 10.3945/jn.115.222620. Epub 2016 Jan 13. PMID 26764319
- [Derived] Sorensen LB, Dyssegaard CB, Damsgaard CT, Petersen RA, Dalskov SM, Hjorth MF, Andersen R, Tetens I, Ritz C, Astrup A, Lauritzen L, Michaelsen KF, Egelund N. The effects of Nordic school meals on concentration and school performance in 8- to 11-year-old children in the OPUS School Meal Study: a cluster-randomised, controlled, cross-over trial. Br J Nutr. 2015 Apr 28;113(8):1280-91. doi: 10.1017/S0007114515000033. Epub 2015 Mar 20. PMID 25791747
- [Derived] Dalskov SM, Ritz C, Larnkjaer A, Damsgaard CT, Petersen RA, Sorensen LB, Ong KK, Astrup A, Molgaard C, Michaelsen KF. The role of leptin and other hormones related to bone metabolism and appetite regulation as determinants of gain in body fat and fat-free mass in 8-11-year-old children. J Clin Endocrinol Metab. 2015 Mar;100(3):1196-205. doi: 10.1210/jc.2014-3706. Epub 2014 Dec 22. PMID 25532044
- [Derived] Hjorth MF, Quist JS, Andersen R, Michaelsen KF, Tetens I, Astrup A, Chaput JP, Sjodin A. Change in sleep duration and proposed dietary risk factors for obesity in Danish school children. Pediatr Obes. 2014 Dec;9(6):e156-9. doi: 10.1111/ijpo.264. Epub 2014 Sep 24. PMID 25251317